CLINICAL TRIAL: NCT07338942
Title: A Prospective, Multicenter, Intervention Study to Evaluate the Impact of the Implementation of Standardized Transthyretin Amyloidosis (ATTR) Early Identification and Diagnosis in ATTR High Risk Population
Brief Title: Implementation of Standardized Early Identification and Diagnosis for Transthyretin Amyloidosis (ATTR) in High-Risk Populations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D8455L00002
Record Dates: First submitted 2025-12-03; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: ATTR-CM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm without control group (Other): This is a multi-center, prospective, single-arm interventional study to evaluate the impact of the implementation of standardized ATTR early identification and diagnosis in ATTR high risk population. This study will enroll approximately 4,000 adult Chinese patients at high risk for ATTR from around 50 sites in China.
  Interventions: Behavioral: implementation of standard early identification and diagnosis of ATTR

INTERVENTIONS:
Behavioral: implementation of standard early identification and diagnosis of ATTR — The intervention methods include standardized ATTR early identification and diagnosis protocol, as well as quality audit.
  The standardized ATTR early identification and diagnosis protocol involves knowledge training, operation training and verification.

SUMMARY:
This multicenter, prospective, single-arm, interventional study will enroll about 4,000 adult patients at high risk of ATTR amyloidosis from around 50 sites in China. Eligible patients are aged ≥60 years and have documented symptomatic heart failure with left ventricular ejection fraction ≥40% and LVH. Exclusion criteria include known etiologies of myocardial diseases, anomalies of serum free light chain or serum immunofixation electrophoresis, acute myocardial infarction within 6 months before screening, and inability to undergo 99mTc-PYP. Patients will undergo a 14-week diagnostic process.

The study intervention involves knowledge training, operation training and post-training verification among investigators. Knowledge training for CV department investigators will cover disease-specific knowledge, standard diagnostic pathways, and genetics; training for investigators in echocardiology (ECHO) and nuclear medicine departments will focus on disease knowledge, standardized operating procedures (SOPs), and imaging parameter reporting. Operation training includes hands-on training in SOPs and image interpretation for ECHO and nuclear medicine investigators. Post-training verification will assess site-level compliance. Extra training will be arranged if quality audit is off target.

The primary endpoint is the proportion of patients diagnosed with ATTR amyloidosis in high-risk populations. Secondary endpoints include the proportion of patients with ATTRwt amyloidosis, concordance between local investigators and central reviewers in ECHO and 99mTc-PYP readings, and genotype distribution. All analyses will be descriptive with no pre-planned hypotheses. Risk factors associated with 99mTc-PYP-diagnosed ATTR amyloidosis will be analyzed via logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years, at the time of signing the informed consent (ICF).
2. Documented diagnosis of symptomatic heart failure (NYHA class I-III) at enrolment, and current diagnosis or a medical history of HF
3. Documented Elevated N-terminal pro-B-type natriuretic peptide (NT-proBNP) > 300 pg/mL at enrolment.
4. Documented LVEF ≥40% at enrolment.
5. Documented LVH defined as end-diastolic wall thickness of ≥12 mm (IVS or PWT) on transthoracic Echocardiogram (TTE) at enrolment.
6. Patients who are willing and able to comply with all scheduled visits, laboratory tests, and other study procedures.
7. Willing and able to undergo 99mTc-PYP scintigraphy.
8. Capable of giving signed ICF as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Known etiology of myocardial disease: A confirmed diagnosis of amyloidosis (e.g., amyloid A amyloidosis, primary [light chain] amyloidosis), a non-amyloid infiltrative cardiomyopathy (i.e., cardiac sarcoidosis, hemochromatosis), muscular dystrophies, cardiomyopathy with reversible causes, hypertensive heart disease, pheochromocytoma, hypertrophic obstructive cardiomyopathy with known geneticetiology, or known pericardial constriction, etc. These diagnoses of myocardial disease could be further validated by the Investigator at Screening if the prior diagnosis is considered suspect.
2. Known serum free light chain (sFLC), serum immunofixation electrophoresis (sIFE), or urine immunofixation electrophoresis (uIFE) anomalies.
3. Prior clinical history of Coronary Artery Bypass Grafting (CABG) or multi-vessel obstructive coronary disease (>50% stenosis of >2 epicardial coronary arteries).
4. Acute Myocardial Infarction (AMI) within 6 months before Screening.
5. Unable to undergo 99mTc-PYP examination, such as:

1)Previously documented hypersensitivity reaction to 99mTc; 2)Severe renal insufficiency (eGFR <30 mL/min/1.73m²); 3)Severe myelosuppression (leukocytes <3.5×10⁹/L or platelets <80×10⁹/L). 6.Other medical or psychiatric condition including recent (within the past year) active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the patient inappropriate for the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with ATTR in high-risk population. | Week 14

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Zhongshan Hospital, Shanghai, Shanghai Municipality, China